CLINICAL TRIAL: NCT01131793
Title: Total Occlusion With Angioplasty After Using a Radiofrequency Guide Wire-Magnetic-Coronary
Brief Title: PowerAssert Radio-Frequency (RF) Guidewire Coronary In-Stent Chronic Total Occlusion (CTO)
Acronym: TOTAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stereotaxis (Industry)
Responsible Party: Mark Jacob, Stereotaxis Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-019
Record Dates: First submitted 2010-05-20; First posted 2010-05-27 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Chronic Total Occlusion In-Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF Guidewire (Experimental)
  Interventions: Device: PowerAssert RF wire in crossing coronary in-stent chronic total occlusions

INTERVENTIONS:
Device: PowerAssert RF wire in crossing coronary in-stent chronic total occlusions — Radio frequency ablation of chronic total occlusions within a stent of a coronary artery using Niobe Magnetic Navigation System (MNS) and the PowerAssert Radiofrequency Guidewire
  Other Names: PowerAssert RF; Magnetic RF Wire

SUMMARY:
A single center Pilot Clinical Registry Study of the" Acute Procedural" Safety and Efficacy of Stereotaxis PowerAssert(TM)RF Coronary Total Occlusion System assisted Angioplasty in the Treatment of Refractory Coronary Total Occlusions

DETAILED DESCRIPTION:
Determine the safety and efficacy of the Stereotaxis PowerAssert™ 18 RF Wire System:

Primary - of recanalizing (crossing) coronary total occlusions within a stent.

Secondary - facilitated angioplasty at hospital discharge represented by

* Event free survival
* Anginal status, and
* Target vessel patency
* minimal luminal diameter (MLD).

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for elective revascularization of a native coronary vessel
* Patient has refractory coronary total occlusion (Thrombolysis In Myocardial Infarction (TIMI) 0 flow) within a stent
* Written Informed Consent obtained

Exclusion Criteria:

* Under 18 years of age
* Current participation in another study with any investigational drug or device

  ->TIMI 0 flow at target lesion site
* Lesion >40mm. in length
* Factors making follow-up or repeat angiography difficult or unlikely
* Acute myocardial infarction less than 1 month before angioplasty
* Contra-indication to emergency coronary artery bypass surgery
* No access to cardiac surgery
* Contra-indication to treatment with aspirin, ticlopidine, clopidogrel or heparin
* Angiographic evidence of thrombus (filling defect proximal to or involving the occlusion)
* Occluded ostium of the right coronary artery or stem of left main coronary artery as target lesion
* Totally occluded bypass graft as target vessel
* Occlusion in an unprotected left main coronary artery
* Ejection fraction less than 30%
* Lesion beyond acute bends or in a location within the coronary anatomy where the catheter cannot traverse
* Lesion within a bifurcation with a significant sidebranch >1.5mm in diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Primary RF wire success | Assessed and measured during interventional procedure up to discharge-average hospital stay 1-5 days- defined in protocol as the number of days between interventional treatment and hospital discharge
  Defined as reaching the true lumen of any branch distal to the total occlusion with the sole use of the RF wire with absence of major complications (Myocardial Infarction (MI), tamponade, emergency Cornary Artery Bypass graft (CABG) or death)

SECONDARY OUTCOMES:
Facilitated RF wire Success: Procedure Success: Clinical Success | Assessed and measured during interventional procedure up to discharge-average hospital stay 1-5 days- defined in protocol as the number of days between interventional treatment and hospital discharge
  Facilitated RF wire success is defined as reaching the true lumen of any branch distal to the total occlusion with combined use of the RF wire and any approved mechanical guidewire with absence of major complications Procedure success defined as in-hospital device success and final residual stenosis < 30% on visual assessment, following adjunctive angioplasty, with absence of major complications Clinical success defined as device and procedure success during the concurrent hospital stay with absence of major complication

CONTACTS AND LOCATIONS:
Overall Officials: Projessor Patrick W. Serruys, PhD, Principal Investigator — Erasmus Medical University Thoraxcenter
Locations (1):
- Erasmus MC University Medical Center, Rotterdam, The Netherlands, Netherlands